CLINICAL TRIAL: NCT00662025
Title: A Phase II Study Of Sunitinib Malate In Combination With Capecitabine In Patients With Advanced Or Metastatic Breast Cancer
Brief Title: Study Of Sunitinib With Capecitabine In Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181163
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2010-10-13 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Advanced/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Capecitabine; Drug: Sunitinib

INTERVENTIONS:
Drug: Capecitabine — Capecitabine 1000 mg/m2, twice daily, for 2 consecutive weeks, followed by a 1-week rest period and given as 3-week cycles
Drug: Sunitinib — Sunitinib 37.5 mg daily, continuous dosing

SUMMARY:
To evaluate efficacy, safety and pharmacokinetics of sunitinib plus Capecitabine in Japanese patients with advanced/metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-proven diagnosis of breast adenocarcinoma that is not amenable to surgery, radiation, or combined modality therapy with curative intent
* Measurable disease as per RECIST. Measurable lesions that have been previously irradiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy.
* Prior treatment with an anthracycline and a taxane in the neoadjuvant, adjuvant or metastatic disease settings.

Exclusion Criteria:

* Histology of inflammatory carcinoma with no other measurable disease. Patients with histology of inflammatory carcinoma are allowed on study if they have measurable disease.
* Brain metastases, spinal cord compression, or carcinomatous meningitis, or leptomeningeal disease.
* Prior treatment with 5-fluorouracil (5-FU) and 5-FU derivatives such as Furtulon (5'-DFUR), Futraful/ Sunfural (tegafur), UFT/UFT-E (tegafur/uracil), TS-1 (tegafur/gimeracil/oteracil) or Mifurol (carmofur) in metastatic disease setting

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- Japan (17):
  - Pfizer Investigational Site, Anjo, Aichi-ken
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Okazaki, Aichi-ken
  - Pfizer Investigational Site, Toyoake, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Morioka, Iwate
  - Pfizer Investigational Site, Kyoto, Japan
  - Pfizer Investigational Site, Kagoshima, Kagoshima-ken
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Osaka, Osaka
  - Pfizer Investigational Site, Sakai, Osaka
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Koto-ku, Tokyo
  - Pfizer Investigational Site, Niigata

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181163&StudyName=Study%20Of%20Sunitinib%20With%20Capecitabine%20In%20Breast%20Cancer

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 cohorts. Cohort 1 enrolled 6 participants. All adverse events in Cohort 1 were evaluated at the end of Cycle 2, and study continuation to Cohort 2 was determined based on the recommendation from the Independent Safety Monitoring Committee. Cohort 2 consisted of 63 participants, including the 6 participants in Cohort 1.
Groups:
- SUNITINIB+CAPECITABINE: Sunitinib was administered orally from Day 1 at the starting dose of 37.5 mg/day on a continuous daily dosing schedule in 21-day cycles. Capecitabine was administered orally from Days 1 to 14 every 21 days at a starting dose of 2,000 mg/m^2/day. Participants were monitored for toxicity, and sunitinib and/or capecitabine dosing could be interrupted or reduced according to individual tolerance. Participants with progressive disease (PD) or intolerable toxicity were considered for discontinuation from the study.
Period: Overall Study
Arm/Group | SUNITINIB+CAPECITABINE
Started | 63 (All 63 participants were included in Full Analysis Set population.)
Completed | 0
Not Completed | 63
Not completed — Objective progression or relapse | 51
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Results of other clinical study | 2
Not completed — Target lesion cannot be evaluated | 1
Not completed — Domestic circumstances | 1

BASELINE CHARACTERISTICS:
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
Age Continuous [Mean (Full Range); unit: years] | 52.9 [26 to 76]
Age, Customized [Number; unit: participants]
  >=20 years and 44 years >= | 13
  >=45 years and 64 years >= | 43
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63
  Male | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Score 0: Fully active, able to carry on all pre-disease performance without restriction.
  Score 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  participants
    Score 0 | 57
    Score 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Based on Data Review Committee's Assessment
Description: Number of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST). CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the longest dimensions (LDs) of the target lesions taking as reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat evaluation ≥4 weeks after initial documentation of response.
Time Frame: Day 1 of Cycle 2, every 6 weeks after Cycle 2, and at the end of Cycle 8.
Population: Full Analysis Set (FAS) is defined as the population of all participants who are diagnosed as having advanced/metastatic breast cancer and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
participants
  Total Number of Participants with CR+PR | 19
  Complete Response (CR) | 0
  Partial Response (PR) | 19
Statistical Analysis 1: Comparison: SUNITINIB+CAPECITABINE; Test type: Superiority or Other; Objective Response Rate (percentage) = 30.2, 95% CI 2-sided [19.2 to 43.0]

2. Secondary Outcome: Number of Participants With Objective Response Based on Investigator's Assessment
Description: Number of participants with objective response based on assessment of confirmed CR or confirmed PR according to RECIST. CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the LDs of the target lesions taking as reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat evaluation ≥4 weeks after initial documentation of response.
Time Frame: Day 1 of Cycle 2, every 6 weeks after Cycle 2, and at the end of study.
Population: FAS is defined as the population of all participants who are diagnosed as having advanced/metastatic breast cancer and received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
participants
  Total Number of Participants with CR+PR | 17
  Complete Response (CR) | 0
  Partial Response (PR) | 17
Statistical Analysis 1: Comparison: SUNITINIB+CAPECITABINE; Test type: Superiority or Other; Objective Response Rate (percentage) = 27.0, 95% CI 2-sided [16.6 to 39.7]

3. Secondary Outcome: Number of Participants With Clinical Benefit Response (CBR) Based on Data Review Committee's Assessment
Description: Number of participants with confirmed CR, PR or stable disease (SD) for at least 24 weeks on study according to RECIST. CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the LDs of the target lesions taking as a reference the baseline sum LD according to RECIST. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of LDs since treatment started.
Time Frame: Day 1 of Cycle 2, every 6 weeks after Cycle 2, and at the end of Cycle 8.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
participants
  Total Number of Participants with CBR | 32
  Complete Response (CR) | 0
  Partial Response (PR) | 19
  Stable Disease (SD) >= 168 days | 13
Statistical Analysis 1: Comparison: SUNITINIB+CAPECITABINE; Test type: Superiority or Other; CBR Rate (percentage) = 50.8, 95% CI 2-sided [37.9 to 63.6]

4. Secondary Outcome: Number of Subjects With CBR Based on Investigator's Assessment
Description: Number of participants with confirmed CR, PR or SD for at least 24 weeks on study according to RECIST. CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the LDs of the target lesions taking as a reference the baseline sum LD according to RECIST. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as reference smallest sum of LDs since treatment started.
Time Frame: Day 1 of Cycle 2, every 6 weeks after Cycle 2, and at the end of study.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
participants
  Total Number of Participatnts with CBR | 33
  Complete Response (CR) | 0
  Partial Response (PR) | 17
  Stable Disease (SD) >= 168 days | 16
Statistical Analysis 1: Comparison: SUNITINIB+CAPECITABINE; Test type: Superiority or Other; CBR Rate (percentage) = 52.4, 95% CI 2-sided [39.4 to 65.1]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Based on Data Review Committee's Assessment. PFS is defined as the time from the start of study treatment to first documentation of objective tumor progression, or to death on study due to any cause, whichever occurred first.
Time Frame: Day 1 of Cycle 2, every 6 weeks after Cycle 2, and at the end of Cycle 8. Up to 28 days after the last administration of the study drug.
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
months | 5.3 [4.1 to 5.7]

6. Secondary Outcome: Time to Tumor Progression (TTP)
Description: Based on Data Review Committee's Assessment. TTP is defined as the time from the start of study treatment to first documentation of objective tumor progression.
Time Frame: as for outcome 5
Population: FAS is defined as the population of all enrolled patients who are diagnosed as having advanced/metastatic breast cancer and received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
months | 5.3 [4.1 to 5.7]

7. Secondary Outcome: Duration of Objective Tumor Response (DR)
Description: Based on Data Review Committee's Assessment. DR is defined as the time from the first documentation of objective tumor response (confirmed CR or PR) to the first documentation of disease progression or to death due to cancer, whichever occurred first. CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the LDs of the target lesions taking as reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat evaluation ≥4 weeks after initial documentation of response.
Time Frame: as for outcome 5
Population: FAS is defined as the population of all participants who are diagnosed as having advanced/metastatic breast cancer and received at least one dose of study medication.
  Nineteen participants with objective tumor response were analyzed for DR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 19
months | 4.1 [2.8 to 5.4]

8. Secondary Outcome: Time to Objective Tumor Response (TTR)
Description: Based on Data Review Committee's Assessment. TTR is defined as the time from the start of study treatment to first documentation of objective tumor response (confirmed CR or PR). CR is defined as disappearance of all target and non-target lesions. PR is defined as ≥30% decrease in sum of the LDs of the target lesions taking as reference the baseline sum LD according to RECIST. Confirmed responses are those that persist on repeat evaluation ≥4 weeks after initial documentation of response.
Time Frame: as for outcome 5
Population: FAS is defined as the population of all participants who are diagnosed as having advanced/metastatic breast cancer and received at least one dose of study medication.
  Twenty three participants with objective tumor response were analyzed for TTR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 23
months | 1.4 [1.3 to 1.4]

9. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the start of study treatment to death due to any cause. OS data is censored on the last day they were known to be alive in the absence of confirmation of death.
Time Frame: A survival survey was conducted at least every 6 months after the completion of study treatment or withdrawal from the study.
Population: as for outcome 2
Measure: Median (Full Range); unit: months
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 63
months | 20.0 [17.2 to NA] — The upper confidence interval was not calculated due to immature follow-up data.

10. Secondary Outcome: Trough Plasma Concentration (Ctrough) for Sunitinib, SU012662, and Total Drug (Sunitinib+SU012662)
Description: SU012662 is a metabolite of sunitinib. Trough plasma concentration (Ctrough) means the concentration prior to study drug administration.
  The Ctrough for total drug (sunitinib+SU012662) was calculated as the mean of the Ctrough of total drug from individual participant.
Time Frame: Days 14 and 15 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants (Cohort 1).
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
nanogram/milliliter
  Sunitinib | 68.7 (16.7)
  SU012662 | 30.8 (10.2)
  Total Drug (Sunitinib+SU012662) | 99.5 (24.1)

11. Secondary Outcome: Tmax for Sunitinib, SU012662, and Total Drug (Sunitinib+SU012662)
Description: SU012662 is a metabolite of sunitinib. Tmax means a time to first occurrence of maximum observed plasma concentration (Cmax).
  The Tmax for total drug (sunitinib+SU012662) was calculated as the median of the Tmax of total drug from individual participant.
Time Frame: Days 14 and 15 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants (Cohort 1).
Measure: Median (Full Range); unit: hours
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
hours
  Sunitinib | 10 [6 to 24]
  SU012662 | 3 [0 to 10]
  Total Drug (Sunitinib+SU012662) | 6 [0 to 10]

12. Secondary Outcome: Cmax for Sunitinib, SU012662, and Total Drug (Sunitinib+SU012662)
Description: SU012662 is a metabolite of sunitinib. Cmax means a maximum observed plasma concentration.
  The Cmax for total drug (sunitinib+SU012662) was calculated as the mean of the Cmax of total drug from individual participant.
Time Frame: Days 14 and 15 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants (Cohort 1).
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
nanogram/milliliter
  Sunitinib | 87.7 (27.6)
  SU012662 | 33.9 (8.43)
  Total Drug (Sunitinib+SU012662) | 119 (31.7)

13. Secondary Outcome: AUC(0-24) for Sunitinib, SU012662, and Total Drug (Sunitinib+SU012662)
Description: SU012662 is a metabolite of sunitinib. AUC(0-24) means an area under the plasma concentration time curve from time zero to 24 hours post-dose.
  The AUC(0-24) for total drug (sunitinib+SU012662) was calculated as the mean of the AUC(0-24) of total drug from individual participant.
Time Frame: Days 14 and 15 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants (Cohort 1).
Measure: Mean (Standard Deviation); unit: nanogram∙hour/milliliter
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
nanogram∙hour/milliliter
  Sunitinib | 1886 (524)
  SU012662 | 704 (176)
  Total drug (Sunitinib+SU012662) | 2590 (658)

14. Secondary Outcome: Tmax for Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR and 5-FU)
Description: Tmax means a time to first occurrence of maximum observed plasma concentration (Cmax).
  5'-DFCR = 5'-deoxy-5-fluorocytidine, 5'-DFUR = 5'-deoxy-5-fluorouridine, 5-FU = 5-fluorouracil
Time Frame: Day 14 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants (Cohort 1).
  n=Number of participants with analyzable data.
Measure: Median (Full Range); unit: hours
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
hours
  Capecitabine (n=4) | 0.75 [0.5 to 2]
  5'-DFCR (n=4) | 1 [1 to 2]
  5'-DFUR (n=4) | 1.5 [1 to 2]
  5-FU (n=4) | 1.5 [1 to 2]

15. Secondary Outcome: Cmax for Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR and 5-FU)
Description: Cmax means a maximum observed plasma concentration. 5'-DFCR = 5'-deoxy-5-fluorocytidine, 5'-DFUR = 5'-deoxy-5-fluorouridine, 5-FU = 5-fluorouracil
Time Frame: Day 14 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 subjects (Cohort 1). n=Number of subjects with analyzable data.
Measure: Mean (Standard Deviation); unit: nanogram/milliliter
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
nanogram/milliliter
  Capecitabine (n=4) | 3773 (1907)
  5'-DFCR (n=4) | 5758 (2405)
  5'-DFUR (n=4) | 6885 (4130)
  5-FU (n=4) | 387 (249)

16. Secondary Outcome: AUC(0-inf) for Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR and 5-FU)
Description: AUC(0-inf) means an area under the plasma concentration time curve from time zero to Infinity.
  5'-DFCR = 5'-deoxy-5-fluorocytidine, 5'-DFUR = 5'-deoxy-5-fluorouridine, 5-FU = 5-fluorouracil
Time Frame: Day 14 of Cycle 1
Population: Pharmacokinetic parameters are estimated for the initial 6 participants(Cohort 1).
  n=Number of participants with analyzable data.
Measure: Mean (Standard Deviation); unit: nanogram∙hour/milliliter
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
nanogram∙hour/milliliter
  Capecitabine (n=3) | 5505 (151)
  5'-DFCR (n=4) | 13177 (7038)
  5'-DFUR (n=3) | 12236 (3777)
  5-FU (n=3) | 635 (152)

17. Secondary Outcome: t1/2 for Capecitabine and Its Metabolites (5'-DFCR, 5'-DFUR and 5-FU)
Description: t1/2 means a terminal phase half-life. 5'-DFCR = 5'-deoxy-5-fluorocytidine, 5'-DFUR = 5'-deoxy-5-fluorouridine, 5-FU = 5-fluorouracil
Time Frame: Day 14 of Cycle 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | SUNITINIB+CAPECITABINE
Number analyzed (Participants) | 6
hours
  Capecitabine (n=3) | 0.80 (0.34)
  5'-DFCR (n=4) | 1.01 (0.19)
  5'-DFUR (n=3) | 0.73 (0.05)
  5-FU (n=3) | 0.77 (0.06)

ADVERSE EVENTS:
Time Frame: Up to 28 days after the last administration of the study drug
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | SUNITINIB+CAPECITABINE
Serious Adverse Events (participants affected / at risk) | 17/63
Other Adverse Events (participants affected / at risk) | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SUNITINIB+CAPECITABINE (N=63)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Ascites (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gingival bleeding (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Malaise (General disorders) | 2
Pyrexia (General disorders) | 2
Hepatic function abnormal (Hepatobiliary disorders) | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SUNITINIB+CAPECITABINE (N=63)
Anaemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 46
Lymphopenia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 59
Thrombocytopenia (Blood and lymphatic system disorders) | 58
Hyperthyroidism (Endocrine disorders) | 6
Hypothyroidism (Endocrine disorders) | 15
Dry eye (Eye disorders) | 4
Eyelid oedema (Eye disorders) | 13
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 12
Cheilitis (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 16
Diarrhoea (Gastrointestinal disorders) | 35
Dry mouth (Gastrointestinal disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 8
Gingival bleeding (Gastrointestinal disorders) | 5
Gingivitis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 38
Stomatitis (Gastrointestinal disorders) | 30
Vomiting (Gastrointestinal disorders) | 28
Chills (General disorders) | 4
Face oedema (General disorders) | 18
Fatigue (General disorders) | 39
Mucosal inflammation (General disorders) | 5
Oedema (General disorders) | 5
Oedema peripheral (General disorders) | 15
Pyrexia (General disorders) | 20
Hepatic function abnormal (Hepatobiliary disorders) | 19
Nasopharyngitis (Infections and infestations) | 15
Urinary tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 10
Aspartate aminotransferase increased (Investigations) | 12
Blood bilirubin increased (Investigations) | 7
Blood lactate dehydrogenase increased (Investigations) | 7
Blood thyroid stimulating hormone increased (Investigations) | 13
Blood urine present (Investigations) | 6
Ejection fraction decreased (Investigations) | 7
Haemoglobin decreased (Investigations) | 9
Weight decreased (Investigations) | 17
Hypoalbuminaemia (Metabolism and nutrition disorders) | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 36
Headache (Nervous system disorders) | 17
Insomnia (Psychiatric disorders) | 8
Proteinuria (Renal and urinary disorders) | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 4
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 5
Nail disorder (Skin and subcutaneous tissue disorders) | 8
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 45
Rash (Skin and subcutaneous tissue disorders) | 18
Skin discolouration (Skin and subcutaneous tissue disorders) | 13
Haemorrhage (Vascular disorders) | 5
Hypertension (Vascular disorders) | 18
Blood phosphorus decreased (Investigations) | 4
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Hypoaesthesia (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.